CLINICAL TRIAL: NCT00172367
Title: Chemoprevention Trial for Uremia-Associated Urothelial Carcinoma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: This study was for National Science Council project. The study was not funded, so the study was withdrawn.
Sponsor: National Taiwan University Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 930906
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2008-09-26 (Estimated); Status verified 2004-11

CONDITIONS: Carcinoma, Transitional Cell
Keywords: Urothelial carcinoma; Lycopene; uremia; prevention; biomarker; progression; anti-oxidant
MeSH Terms: conditions — Carcinoma, Transitional Cell; Uremia; Disease Progression | interventions — Lycopene

INTERVENTIONS:
Drug: Lycopene

SUMMARY:
Primary Objective: To study if lycopene can improve the biomarker status of urothelial cells in patients with uremia-associated urothelial carcinoma.

Secondary Objective: To evaluate the general safety and tolerability of oral lycopene 30 mg per day for 12 weeks in uremic patients.

DETAILED DESCRIPTION:
This is a renal function-stratified phase II chemoprevention trial. After 8 weeks of a run-in and washout period, participants will take lycopene, 30 mg per day for 12 weeks. The expression of intermediate biomarkers will be determined upon study entry after 8 weeks of run-in/washout, and after 6 and 12 weeks of lycopene supplementation. It takes at least 20 weeks to complete the course.

ELIGIBILITY:
Inclusion Criteria:

* Patients have pathologically-proven urothelial carcinoma (UC) with a clinical stage <= T3N0M0
* Patients have no visible or identifiable residual UC after treatment with a life expectancy of > 6 months
* Patients have remaining urothelium at risk of recurrence (transplanted renal unit excluded)
* No other active malignancy. Patients who have other primary malignancies should be treated successfully prior to the study entry and should be in a cure or remission state for at least one year.
* Patients are able to take lycopene capsules orally.
* Patients who sign and give informed consents and are willing to conform to the scheduled sampling of the blood, urine and/or tissue

Exclusion Criteria:

* Patients who have clinical stage > T3N0M0 or metastatic disease
* Positive urine cytology. Patients who have positive cytology should be subjected to a serial diagnostic workup which may include renal echo, cystoscopy and ureterorenoscopy, and image studies (intravenous urography, computed tomography, magnetic resonance urography, retrograde or antegrade pyelography). If no recurrent or residual tumors are found, patients are still eligible for the study.
* Patients who have ever received systemic chemotherapy within 12 months
* Patients who have gastrointestinal malabsorption regardless of the etiology
* Have known allergic reaction to tomato or lycopene
* Patients who are participating or will participate in other clinical trials
* Patients who have active urinary tract infection can not be accrued until infection is effectively controlled
* Patient's age is less than 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2006-01

PRIMARY OUTCOMES:
changes of intermediate biomarker status after lycopene supplementation

SECONDARY OUTCOMES:
safety and tolerability

CONTACTS AND LOCATIONS:
Overall Officials: Yeong-Shiau Pu, MD, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan